CLINICAL TRIAL: NCT00891176
Title: Persistence of Antibodies After Full Vaccination Course With GSK Biologicals' Menitorix or MenC Conjugate Vaccine, Co-administered With DTPa or DTPa/Hib Containing Vaccine and Pneumococcal Conjugate Vaccine, in Children up to 6 Years of Age
Brief Title: Persistence of Antibodies at 3, 4 and 6 Years of Age After Vaccination With Meningococcal, Pneumococcal and Hib Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112830
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-09

CONDITIONS: Neisseria Meningitidis; Haemophilus Influenzae Type b
Keywords: Conjugate vaccines; Meningococcal serogroup C vaccine; Antibody persistence; Pneumococcal vaccine; Haemophilus Influenzae type b vaccine
MeSH Terms: conditions — Haemophilus Infections

ARMS (4):
- Synflorix-Meningitec Group (Experimental): Subjects who received concomitantly in the primary study (NCT00334334): 3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age 2 primary doses of Meningitec intramuscularly into the lower left thigh at 2 and 4 months of age. 3 primary doses of Infanrix hexa intramuscularly into the upper left thigh at 2, 4 and 6 months of age. (In Poland subjects were offered a third dose of Meningitec at 7 months of age to comply with national recommendations). During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV/Hib was given instead of Infanrix hexa.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: MeningitecTM; Biological: InfanrixTM hexa; Biological: InfanrixTM IPV/Hib
- Synflorix-NeisVac-C Group (Experimental): Subjects who received concomitantly in the primary study (NCT00334334): 3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age, 2 primary doses of Neis-Vac-C intramuscularly into the lower left thigh at 2 and 4 months of age and 3 primary doses of Infanrix hexa intramuscularly into the upper left thigh at 2, 4 and 6 months of age. (In Poland subjects were offered a third dose of Neis-Vac-C at 7 months of age to comply with national recommendations). During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV/Hib was given instead of Infanrix hexa.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: NeisVac-CTM; Biological: InfanrixTM hexa; Biological: InfanrixTM IPV/Hib
- Synflorix-Menitorix Group (Experimental): Subjects who received concomitantly in the primary study (NCT00334334): 3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age, 3 primary doses of Menitorix intramuscularly into the lower left thigh at 2, 4 and 6 months of age and 3 primary doses of Infanrix penta intramuscularly into the upper left thigh at 2, 4 and 6 months of age. During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV was given instead of Infanrix penta.
  Interventions: Biological: MenitorixTM; Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: InfanrixTM penta; Biological: InfanrixTM IPV
- Prevenar-Menitorix Group (Active Comparator): Subjects who received concomitantly in the primary study (NCT00334334): 3 primary doses of Prevenar intramuscularly into the right thigh at 2, 4 and 6 months of age, 3 primary doses of Menitorix intramuscularly into the lower left thigh at 2, 4 and 6 months of age and 3 primary doses of Infanrix penta intramuscularly into the upper left thigh at 2, 4 and 6 months of age. During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV was given instead of Infanrix penta.
  Interventions: Biological: MenitorixTM; Biological: Pneumococcal conjugate vaccine GSK1024850A; Biological: PrevenarTM; Biological: InfanrixTM penta; Biological: InfanrixTM IPV

INTERVENTIONS:
Biological: MenitorixTM — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age and as booster dose at 11-18 months of age. No vaccine was administered during this long-term follow up study.
  Arms: Prevenar-Menitorix Group; Synflorix-Menitorix Group
Biological: Pneumococcal conjugate vaccine GSK1024850A — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age and as booster dose at 11-18 months of age. No vaccine was administered during this long-term follow up study.
Biological: PrevenarTM — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age and as booster dose at 11-18 months of age. No vaccine was administered during this long-term follow up study.
  Arms: Prevenar-Menitorix Group
Biological: MeningitecTM — Intramuscular injection into the thigh as primary vaccination at 2 and 4 months of age and as booster dose at 11-18 months of age. No vaccine was administered during this long-term follow up study
  Arms: Synflorix-Meningitec Group
Biological: NeisVac-CTM — Intramuscular injection into the thigh as primary vaccination at 2 and 4 months of age and as booster dose at 11-18 months of age. No vaccine was administered during this long-term follow up study
  Arms: Synflorix-NeisVac-C Group
Biological: InfanrixTM hexa — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age (all countries) and as booster dose at 11-18 months of age (Germany and Poland). No vaccine was administered during this long-term follow up study
  Arms: Synflorix-Meningitec Group; Synflorix-NeisVac-C Group
Biological: InfanrixTM penta — Intramuscular injection into the thigh as primary vaccination at 2, 4 and 6 months of age (all countries) and as booster dose at 11-18 months of age (Germany and Poland). No vaccine was administered during this long-term follow up study
  Arms: Prevenar-Menitorix Group; Synflorix-Menitorix Group
Biological: InfanrixTM IPV/Hib — Intramuscular injection into the thigh as booster dose at 11-18 months of age (Spain). No vaccine was administered during this long-term follow up study
  Arms: Synflorix-Meningitec Group; Synflorix-NeisVac-C Group
Biological: InfanrixTM IPV — Intramuscular injection into the thigh as booster dose at 11-18 months of age (Spain). No vaccine was administered during this long-term follow up study
  Arms: Prevenar-Menitorix Group; Synflorix-Menitorix Group

SUMMARY:
This protocol posting deals with objectives & outcome measures of an extension phase when subjects are aged 3, 4 and 6 years of age. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00334334). The objectives & outcome measures of the booster phase are presented in a separate protocol posting (NCT number = NCT00463437).

The purpose of this study is to evaluate the persistence of pneumococcal, meningococcal serogroup C, Hib and Hepatits B antibodies after booster vaccination, when the subjects are aged 3, 4 and 6 years. No vaccine will be administered during this persistence phase of the study.

DETAILED DESCRIPTION:
This multicenter study is open. No vaccine will be administered during this persistence phase of the study. The subjects were randomized in the primary vaccination study 107005 and will not be further randomized in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 36 and 40 months of age at the time of Visit 1; between, and including, 48 and 52 months of age at the time of Visit 2; and between, and including, 72 and 76 months of age at the time of Visit 3.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who previously participated in the primary and booster studies, who received a full vaccination course with the vaccines corresponding to their group during the primary and booster studies and who were part, in the booster study, of the blood sampling subset.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first blood sampling.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of any additional meningococcal serogroup C, Hib, hepatitis B and pneumococcal vaccine since the end of the booster study
* History of meningococcal serogroup C, Haemophilus influenzae type b, hepatitis B and invasive pneumococcal diseases since the end of booster study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition since the end of booster study, based on medical history and physical examination (no laboratory testing required).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first blood sampling.

Ages: 36 Months to 76 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 582 (Actual)
Dates: Start 2009-05-14; Primary Completion 2012-11-21 (Actual); Study Completion 2012-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- Germany (21):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oberstenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Tettnang, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Porta Westfalica, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Weimar, Thuringia
  - GSK Investigational Site, Berlin
- Poland (3):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Siemianowice Śląskie
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tejedor JC, Brzostek J, Konior R, Grunert D, Kolhe D, Baine Y, Van Der Wielen M. Antibody Persistence in Young Children 5 Years after Vaccination with a Combined Haemophilus influenzae Type b-Neisseria meningitidis Serogroup C Conjugate Vaccine Coadministered with Diphtheria-Tetanus-Acellular Pertussis-Based and Pneumococcal Conjugate Vaccines. Clin Vaccine Immunol. 2016 Jul 5;23(7):555-63. doi: 10.1128/CVI.00057-16. Print 2016 Jul. PMID 27145999
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112830 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At 3 years of age, 582 subjects were enrolled. One subject who did not participate in the primary study was enrolled by mistake and was therefore withdrawn from the study. Therefore the total number of subjects participating at the 36 months of age time point was 581.
Period: At 3 Years of Age
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Started | 144 | 147 | 149 | 141
Completed | 144 | 147 | 149 | 141
Not Completed | 0 | 0 | 0 | 0
Period: At 4 Years of Age
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Started | 140 | 142 | 142 | 137
Completed | 140 | 142 | 142 | 137
Not Completed | 0 | 0 | 0 | 0
Period: At 6 Years of Age
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Started | 131 | 138 | 135 | 135
Completed | 131 | 138 | 135 | 135
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Synflorix-Meningitec Group: Subjects who received concomitantly in the primary study (NCT00334334): 3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age 2 primary doses of Meningitec intramuscularly into the lower left thigh at 2 and 4 months of age and 3 primary doses of Infanrix hexa intramuscularly into the upper left thigh at 2, 4 and 6 months of age. (In Poland subjects were offered a third dose of Meningitec at 7 months of age to comply with national recommendations). During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV/Hib was given instead of Infanrix hexa.
- Total: Total of all reporting groups
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group | Total
Number analyzed (Participants) | 144 | 147 | 149 | 141 | 581
Age, Continuous [Mean (Standard Deviation); unit: Months] | 37.1 (1.17) | 37.2 (1.20) | 37.3 (1.18) | 37.3 (1.28) | 37.2 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 65 | 86 | 71 | 293
  Male | 73 | 82 | 63 | 70 | 288

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Titers Using Rabbit Complement (rSBA-MenC) Equal to or Above Cut-off Value
Description: rSBA-MenC antibody cut-off value assessed was equal to or above 1:8. The rSBA-MenC assay was performed at the Public Health England (PHE) laboratory at 6 years of age while the GSK laboratory was used for testing at 3 and 4 years of age.
Time Frame: At 3 years of age
Population: Analysis was performed on the According-to-Protocol cohort for antibody persistence at 3 years of age, which included all evaluable subjects who had received the full vaccination course in the primary study (NCT00334334) and in the booster study (NCT00463437) and had available results at 3 years of age.
Measure: Number; unit: subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 139 | 146 | 143 | 137
subjects | 120 | 144 | 127 | 113

2. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Titers Using Rabbit Complement (rSBA-MenC) Equal to or Above Cut-off Value
Description: as for outcome 1
Time Frame: At 6 years of age
Population: Analysis was performed on the According-to-Protocol cohort for antibody persistence at 6 years of age, which included all evaluable subjects who had received the full vaccination course in the primary study (NCT00334334) and in the booster study (NCT00463437) and had available results at 6 years of age.
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 128 | 137 | 130 | 134
Subjects | 31 | 55 | 50 | 34

3. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Titers Using Rabbit Complement (rSBA-MenC) Equal to or Above Cut-off Value
Description: as for outcome 1
Time Frame: At 4 years of age
Population: Analysis was performed on the According-to-Protocol cohort for antibody persistence at 4 years of age, which included all evaluable subjects who had received the full vaccination course in the primary study (NCT00334334) and in the booster study (NCT00463437) and had available results at 4 years of age.
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 134 | 137 | 128 | 128
Subjects | 97 | 132 | 108 | 98

4. Secondary Outcome: Number of Subjects With an rSBA-MenC Titer Equal to or Above Cut-off Value
Description: The cut-off value was defined as a titer equal to or above 1:128.
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 139 | 146 | 143 | 137
subjects | 69 | 109 | 98 | 68

5. Secondary Outcome: rSBA-MenC Titers
Description: Titers are given as Geometric Mean Titers (GMTs).
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 139 | 146 | 143 | 137
Titer | 100.5 [75.6 to 133.8] | 235.3 [189.1 to 292.7] | 167.5 [126.0 to 222.7] | 84.0 [61.6 to 114.6]

6. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations Equal to or Above Cut-off Values
Description: The cut-off values were defined as a concentration equal to or above 0.15 microgram per milliliter (μg/mL) and equal to or above 1.0 μg/mL.
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 132 | 139 | 137 | 138
subjects
  ≥ 0.15 µg/mL | 132 | 139 | 137 | 138
  ≥ 1.0 µg/mL | 101 | 105 | 127 | 115

7. Secondary Outcome: Anti-PRP Concentrations
Description: Concentrations were defined as Geometric Mean Concentrations (GMCs) in μg/mL,
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 132 | 139 | 137 | 138
μg/mL | 2.293 [1.870 to 2.812] | 2.222 [1.794 to 2.752] | 4.177 [3.427 to 5.092] | 3.636 [2.957 to 4.471]

8. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: Antibody concentrations were expressed as GMCs in μg/mL.
  Vaccine pneumococcal serotypes assessed included 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 141 | 146 | 144 | 140
μg/mL
  Anti-1 (N= 139; 146; 142; 139) | 0.26 [0.22 to 0.30] | 0.23 [0.19 to 0.26] | 0.21 [0.18 to 0.25] | 0.07 [0.06 to 0.09]
  Anti-4 (N= 141; 146; 144; 139) | 0.27 [0.23 to 0.32] | 0.23 [0.20 to 0.27] | 0.23 [0.20 to 0.27] | 0.35 [0.29 to 0.42]
  Anti-5 (N= 140; 145; 144; 140) | 0.46 [0.39 to 0.54] | 0.39 [0.33 to 0.46] | 0.41 [0.35 to 0.50] | 0.09 [0.07 to 0.10]
  Anti-6B (N= 139; 146; 144; 138) | 0.59 [0.45 to 0.76] | 0.56 [0.45 to 0.71] | 0.63 [0.47 to 0.84] | 0.95 [0.77 to 1.18]
  Anti-7F (N= 141; 146; 144; 140) | 0.58 [0.50 to 0.67] | 0.51 [0.43 to 0.59] | 0.54 [0.45 to 0.66] | 0.07 [0.05 to 0.09]
  Anti-9V (N= 141; 146; 144; 140) | 0.60 [0.49 to 0.73] | 0.54 [0.44 to 0.66] | 0.47 [0.39 to 0.57] | 0.70 [0.57 to 0.85]
  Anti-14 (N= 141; 146; 144; 140) | 1.33 [1.04 to 1.70] | 1.09 [0.88 to 1.35] | 1.00 [0.80 to 1.25] | 1.48 [1.23 to 1.78]
  Anti-18C (N= 141; 146; 143; 139) | 0.60 [0.50 to 0.71] | 0.84 [0.73 to 0.97] | 0.59 [0.48 to 0.71] | 0.59 [0.50 to 0.70]
  Anti-19F (N= 141; 146; 144; 139) | 2.06 [1.58 to 2.69] | 1.63 [1.27 to 2.09] | 1.35 [1.05 to 1.72] | 1.48 [1.07 to 2.05]
  Anti-23F (N= 140; 146; 144; 140) | 0.73 [0.58 to 0.92] | 0.69 [0.55 to 0.88] | 0.62 [0.46 to 0.82] | 1.36 [1.07 to 1.73]

9. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity
Description: Opsonophagocytic activity was measured by a killing-assay. The results were presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay was an opsonic titre of 8.
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 131 | 131 | 131 | 132
Subjects
  Opsono-1 (N= 131; 131; 131; 131) | 30 | 32 | 29 | 14
  Opsono-4 (N= 126; 127; 129; 128) | 54 | 48 | 43 | 77
  Opsono-5 (N= 130; 130; 129; 132) | 73 | 47 | 55 | 5
  Opsono-6B (N= 128; 127; 124; 131) | 84 | 81 | 78 | 115
  Opsono-7F (N= 131; 130; 131; 130) | 128 | 130 | 131 | 126
  Opsono-9V (N= 131; 131; 129; 132) | 127 | 131 | 127 | 124
  Opsono-14 (N= 129; 128; 128; 131) | 110 | 118 | 106 | 112
  Opsono-18C (N= 126; 121; 123; 122) | 51 | 68 | 44 | 48
  Opsono-19F (N= 130; 130; 131; 132) | 105 | 108 | 89 | 91
  Opsono-23F (N= 125; 124; 125; 132) | 106 | 112 | 113 | 129

10. Secondary Outcome: Concentration of Antibodies Against Protein D
Description: Concentrations were expressed as GMCs in enzyme-linked immunosorbent-assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 140 | 145 | 144 | 139
EL.U/mL | 494.6 [414.0 to 591.0] | 444.8 [373.2 to 530.1] | 439.8 [366.4 to 527.9] | 100.3 [87.6 to 114.9]

11. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above Cut-off Values
Description: Cut-off values assessed were defined as equal to or above 10 milli-international units per milliliter (mIU/mL) or equal to or above 100 mIU/mL.
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 107 | 102 | 105 | 102
subjects
  ≥ 10 mIU/mL | 105 | 96 | 102 | 99
  ≥ 100 mIU/mL | 77 | 81 | 74 | 74

12. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were expressed as GMCs in mIU/mL.
Time Frame: At 3 years of age
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 107 | 102 | 105 | 102
mIU/mL | 367.5 [256.8 to 525.9] | 325.7 [228.3 to 464.7] | 288.1 [198.7 to 417.9] | 371.4 [254.1 to 542.8]

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Related = SAE assessed by the investigator as being related to the study procedures.
Time Frame: From last study contact of the study (NCT00463437) at 17-24 months of age until 3 years of age
Population: Analysis was performed on the Total Enrolled cohort at 3 years of age, which included all subjects vaccinated in the booster study (NCT00463437) and who were part of the blood sample subset.
Measure: Number; unit: subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 144 | 147 | 149 | 141
subjects
  SAE(s) | 0 | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0 | 0

14. Secondary Outcome: rSBA-MenC Titers
Description: Titers are given as Geometric Mean Titers (GMTs).
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 134 | 137 | 128 | 128
Titers | 45.3 [33.2 to 61.8] | 146.8 [116.2 to 185.4] | 112.4 [81.8 to 154.6] | 68.1 [48.4 to 95.9]

15. Secondary Outcome: Number of Subjects With an rSBA-MenC Titer Equal to or Above Cut-off Value
Description: rSBA-MenC antibody cut-off value assessed was equal to or above 1:128.
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 134 | 137 | 128 | 128
Subjects | 49 | 79 | 75 | 58

16. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations Equal to or Above Cut-off Values
Description: as for outcome 6
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Number; unit: Subjects
Groups:
- Synflorix-Meningitec Group: Subjects who received concomitantly in the primary study (NCT00334334): 3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age, 2 primary doses of Meningitec intramuscularly into the lower left thigh at 2 and 4 months of age and 3 primary doses of Infanrix hexa intramuscularly into the upper left thigh at 2, 4 and 6 months of age. (In Poland subjects were offered a third dose of Meningitec at 7 months of age to comply with national recommendations). During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV/Hib was given instead of Infanrix hexa.
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 134 | 136 | 130 | 133
Subjects
  ≥ 0.15 µg/mL | 133 | 134 | 130 | 132
  ≥ 1.0 µg/mL | 88 | 85 | 117 | 106

17. Secondary Outcome: Anti-PRP Concentrations
Description: Concentrations were defined as Geometric Mean Concentrations (GMCs) in μg/mL
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 134 | 136 | 130 | 133
μg/mL | 1.767 [1.454 to 2.146] | 1.738 [1.386 to 2.178] | 3.804 [3.092 to 4.679] | 2.805 [2.297 to 3.425]

18. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: as for outcome 8
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 136 | 138 | 133 | 136
μg/mL
  Anti-1 (N=136;138;131;135) | 0.22 [0.19 to 0.27] | 0.21 [0.17 to 0.26] | 0.18 [0.15 to 0.21] | 0.08 [0.07 to 0.10]
  Anti-4 (N=136;138;131;136) | 0.22 [0.19 to 0.26] | 0.21 [0.18 to 0.25] | 0.20 [0.17 to 0.24] | 0.32 [0.27 to 0.39]
  Anti-5 (N=136;138;131;136) | 0.47 [0.37 to 0.59] | 0.36 [0.30 to 0.42] | 0.34 [0.28 to 0.42] | 0.10 [0.08 to 0.11]
  Anti-6B (N=136;138;133;135) | 0.74 [0.53 to 1.01] | 0.65 [0.49 to 0.86] | 0.78 [0.57 to 1.06] | 0.99 [0.76 to 1.29]
  Anti-7F (N=136;138;131;136) | 0.51 [0.41 to 0.63] | 0.44 [0.37 to 0.52] | 0.46 [0.37 to 0.58] | 0.09 [0.07 to 0.12]
  Anti-9V (N=136;137;131;136) | 0.52 [0.42 to 0.65] | 0.61 [0.46 to 0.81] | 0.54 [0.40 to 0.72] | 0.72 [0.57 to 0.91]
  Anti-14 (N=136;138;132;136) | 1.51 [1.18 to 1.92] | 1.57 [1.25 to 1.97] | 1.41 [1.10 to 1.82] | 1.71 [1.38 to 2.12]
  Anti-18C (N=136;138;132;136) | 0.49 [0.41 to 0.59] | 0.81 [0.67 to 0.98] | 0.60 [0.48 to 0.75] | 0.49 [0.40 to 0.59]
  Anti-19F (N=136;138;133;136) | 2.66 [1.92 to 3.67] | 2.36 [1.70 to 3.29] | 2.50 [1.80 to 3.48] | 2.41 [1.78 to 3.25]
  Anti-23F (N=136;138;133;136) | 0.98 [0.71 to 1.35] | 0.84 [0.65 to 1.10] | 0.98 [0.69 to 1.39] | 1.56 [1.16 to 2.09]

19. Secondary Outcome: Number of Subjects With Opsonophagocytic Activity
Description: Opsonophagocytic activity was measured by a killing-assay. The results were presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay was an opsonic titer of 8.
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 131 | 134 | 123 | 128
Subjects
  Opsono-1 (n=131;134;123;128) | 33 | 32 | 20 | 12
  Opsono-4 (N=127;132;118;126) | 49 | 50 | 36 | 72
  Opsono-5 (N=129;132;122;128) | 65 | 46 | 40 | 5
  Opsono-6B (N=128;129;122;126) | 93 | 97 | 101 | 111
  Opsono-7F (N=131;134;123;128) | 131 | 134 | 123 | 126
  Opsono-9V (N=130;132;120;126) | 125 | 130 | 118 | 122
  Opsono-14 (N=126;128;114;121) | 96 | 105 | 95 | 110
  Opsono-18C (N=113;118;113;118) | 34 | 56 | 46 | 45
  Opsono-19F (N=131;133;123;128) | 87 | 88 | 80 | 89
  Opsono-23F (N=129133;119;121) | 98 | 108 | 86 | 111

20. Secondary Outcome: Concentration of Antibodies Against Protein D
Description: Concentrations were expressed as GMCs in enzyme-linked immunosorbent-assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 136 | 138 | 129 | 132
EL.U/mL | 401.1 [338.3 to 475.6] | 387.2 [326.7 to 458.9] | 334.8 [277.7 to 403.7] | 107.9 [94.6 to 123.1]

21. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above Cut-off Values
Description: as for outcome 11
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 95 | 102 | 98 | 98
Subjects
  ≥ 10 mIU/mL | 86 | 93 | 86 | 90
  ≥ 100 mIU/mL | 67 | 72 | 62 | 72

22. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were expressed as GMCs in mIU/mL.
Time Frame: At 4 years of age
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 95 | 102 | 98 | 98
mIU/mL | 273.5 [183.2 to 408.3] | 238.8 [165.6 to 344.3] | 174.6 [114.5 to 266.4] | 284.7 [190.7 to 425.1]

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From last study contact of the study (NCT00463437) at 17-24 months of age until 4 years of age
Population: Analysis was performed on the Total Enrolled cohort at 4 years of age, which included all subjects vaccinated in the booster study (NCT00463437) and who were part of the blood sample subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 140 | 142 | 142 | 137
Subjects
  SAE(s) | 0 | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects With rSBA-MenC Titer Equal to or Above Cut-off Value
Description: rSBA-MenC antibody cut-off value assessed was equal to or above 1:128.
Time Frame: At 6 years of age
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 128 | 137 | 130 | 134
Subjects | 11 | 19 | 15 | 14

25. Secondary Outcome: rSBA-MenC Titers
Description: Titers are given as Geometric Mean Titers (GMTs).
Time Frame: At 6 years of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 128 | 137 | 130 | 134
Titer | 7.2 [5.8 to 8.9] | 11.9 [8.9 to 16.0] | 10.1 [7.9 to 12.9] | 8.5 [6.6 to 11.1]

26. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations Equal to or Above Cut-off Values
Description: The cut-off values were defined as a concentration ≥ 0.15 microgram per milliliter (μg/mL) and ≥ 1.0 μg/mL.
Time Frame: At 6 years of age
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 127 | 134 | 130 | 132
Subjects
  ≥ 0.15 µg/mL | 126 | 132 | 130 | 132
  ≥ 1.0 µg/mL | 85 | 77 | 110 | 100

27. Secondary Outcome: Anti-PRP Concentrations
Description: Concentrations were defined as Geometric Mean Concentrations (GMCs) in μg/mL
Time Frame: At 6 years of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 127 | 134 | 130 | 132
μg/mL | 1.655 [1.339 to 2.045] | 1.647 [1.298 to 2.090] | 2.947 [2.396 to 3.624] | 2.558 [2.065 to 3.168]

28. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: as for outcome 8
Time Frame: At 6 years of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 128 | 137 | 131 | 134
μg/mL
  Anti-1 (N=128;136;130;134) | 0.19 [0.16 to 0.23] | 0.22 [0.17 to 0.27] | 0.20 [0.15 to 0.26] | 0.11 [0.09 to 0.13]
  Anti-4 (N=128;135;130;134) | 0.14 [0.11 to 0.17] | 0.14 [0.11 to 0.17] | 0.12 [0.10 to 0.15] | 0.24 [0.19 to 0.29]
  Anti-5 (N=128;135;130;131) | 0.37 [0.30 to 0.45] | 0.31 [0.26 to 0.37] | 0.30 [0.25 to 0.37] | 0.13 [0.11 to 0.15]
  Anti-6B (N=128;135;131;131) | 1.71 [1.32 to 2.23] | 1.13 [0.87 to 1.48] | 1.28 [1.00 to 1.64] | 1.73 [1.38 to 2.16]
  Anti-7F (N=127;137;130;132) | 0.61 [0.49 to 0.78] | 0.59 [0.46 to 0.74] | 0.64 [0.50 to 0.82] | 0.24 [0.18 to 0.32]
  Anti-9V (N=128;137;131;132) | 0.76 [0.56 to 1.01] | 0.67 [0.51 to 0.88] | 0.57 [0.42 to 0.79] | 0.65 [0.51 to 0.83]
  Anti-14 (N=128;137;130;133) | 2.84 [2.17 to 3.73] | 2.22 [1.72 to 2.86] | 2.81 [2.07 to 3.81] | 2.59 [2.08 to 3.23]
  Anti-18C (N=128;137;130;132) | 0.52 [0.41 to 0.66] | 0.75 [0.60 to 0.94] | 0.56 [0.43 to 0.74] | 0.49 [0.39 to 0.62]
  Anti-19F (N=128;137;130;133) | 3.91 [3.01 to 5.10] | 3.94 [2.99 to 5.20] | 4.24 [3.30 to 5.45] | 3.11 [2.48 to 3.91]
  Anti-23F (N=128;136;130;133) | 1.71 [1.26 to 2.30] | 1.70 [1.27 to 2.26] | 1.41 [1.06 to 1.87] | 2.99 [2.32 to 3.86]

29. Secondary Outcome: Concentration of Antibodies Against Protein D
Description: Concentrations were expressed as GMCs in enzyme-linked immunosorbent-assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At 6 years of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 128 | 137 | 131 | 133
EL.U/mL | 284.7 [239.5 to 338.4] | 278.0 [236.3 to 327.1] | 266.1 [222.2 to 318.8] | 105.2 [92.4 to 119.8]

30. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above Cut-off Values as Measured by ELISA.
Description: as for outcome 11
Time Frame: At 3 and 4 years of age
Population: as for outcome 2
Measure: Number; unit: Subjects
Groups:
- Synflorix-NeisVac-C Group: Subjects who received concomitantly in the primary study (NCT00334334):
  3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age 2 primary doses of Neis-Vac-C intramuscularly into the lower left thigh at 2 and 4 months of age.
  3 primary doses of Infanrix hexa intramuscularly into the upper left thigh at 2, 4 and 6 months of age.
  (In Poland subjects were offered a third dose of Neis-Vac-C at 7 months of age to comply with national recommendations).
  During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV/Hib was given instead of Infanrix hexa.
- Synflorix-Menitorix Group: Subjects who received concomitantly in the primary study (NCT00334334):
  3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age 3 primary doses of Menitorix intramuscularly into the lower left thigh at 2, 4 and 6 months of age.
  3 primary doses of Pediarix intramuscularly into the upper left thigh at 2, 4 and 6 months of age.
  During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV was given instead of Infanrix penta.
- Prevenar-Menitorix Group: Subjects who received concomitantly in the primary study (NCT00334334):
  3 primary doses of Prevenar intramuscularly into the right thigh at 2, 4 and 6 months of age 3 primary doses of Menitorix intramuscularly into the lower left thigh at 2, 4 and 6 months of age.
  3 primary doses of Infanrix penta intramuscularly into the upper left thigh at 2, 4 and 6 months of age.
  During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV was given instead of Infanrix penta.
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 94 | 98 | 94 | 91
Subjects
  ≥ 10 mIU/mL; 3 years (N= 94, 98, 94, 90) | 92 | 92 | 91 | 87
  ≥ 10 mIU/mL; 4 years (N= 87, 94, 91, 91) | 78 | 86 | 79 | 83
  ≥ 100mIU/mL; 3 years (N= 94, 98, 94, 90) | 71 | 79 | 67 | 67
  ≥ 100mIU/mL; 4 years (N= 87, 94, 91, 91) | 61 | 69 | 57 | 67

31. Secondary Outcome: Anti-HBs Antibody Concentrations as Measured by ELISA
Description: Concentrations were expressed as GMCs in mIU/mL.
Time Frame: At 3 and 4 years of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- Synflorix-Menitorix Group: Subjects who received concomitantly in the primary study (NCT00334334):
  3 primary doses of Synflorix intramuscularly into the right thigh at 2, 4 and 6 months of age 3 primary doses of Menitorix intramuscularly into the lower left thigh at 2, 4 and 6 months of age.
  3 primary doses of Infanrix penta intramuscularly into the upper left thigh at 2, 4 and 6 months of age.
  During the booster study (NCT00463437) subjects received the same vaccines as during the primary study at 11-18 months of age, with the exception of Spain, where Infanrix IPV was given instead of Infanrix penta.
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 94 | 98 | 94 | 91
mIU/mL
  anti-HBs; 3 years (N= 94, 98, 94, 90) | 433.8 [296.2 to 635.2] | 332.3 [230.5 to 479.1] | 302.7 [201.7 to 454.3] | 396.5 [263.4 to 596.9]
  anti-HBs; 4 years (N= 87, 94, 91, 91) | 270.5 [177.0 to 413.5] | 263.1 [180.9 to 382.9] | 172.7 [110.4 to 270.1] | 280.2 [183.6 to 427.7]

32. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations Equal to or Above Cut-off Values
Description: Cut-off values assessed were defined as equal to or above (≥) 6.2 milli-international units per milliliter (mIU/mL), 10 mIU/mL and 100 mIU/mL.
  Note: A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL) when tested by Enzyme-Linked Immunosorbent Assay (ELISA). The tables show both the results obtained by ELISA as well as updated results following complete retesting and reanalysis by a Chemiluminescence immunoassay (CLIA). Anti-HBs seroprotection was redefined as CLIA concentration above 10 mIU/mL.
Time Frame: At 3, 4 and 6 years of age
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 122 | 130 | 125 | 128
Subjects
  ≥ 6.2 mIU/mL; 3 years (N=118,130, 122, 119) | 110 | 121 | 110 | 113
  ≥ 6.2 mIU/mL; 4 years (N= 120, 127, 118, 119) | 110 | 113 | 104 | 109
  ≥ 6.2 mIU/mL; 6 years (N=122, 129, 125, 128) | 102 | 108 | 98 | 112
  ≥ 10 mIU/mL; 3 years (N=118,130, 122, 119) | 109 | 118 | 108 | 111
  ≥ 10 mIU/mL; 4 years (N= 120, 127, 118, 119) | 104 | 112 | 100 | 107
  ≥ 10 mIU/mL; 6 years (N=122, 129, 125, 128) | 100 | 103 | 91 | 108
  ≥ 100 mIU/mL; 3 years (N=118,130, 122, 119) | 80 | 84 | 75 | 74
  ≥ 100 mIU/mL; 4 years (N= 120, 127, 118, 119) | 70 | 76 | 60 | 73
  ≥ 100 mIU/mL; 6 years (N=122, 129, 125, 128) | 57 | 62 | 45 | 66

33. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were expressed as GMCs in mIU/mL. Note: A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL) when tested by ELISA. The tables show both the results obtained by ELISA as well as updated results following complete retesting and reanalysis by a Chemiluminescence immunoassay (CLIA).
Time Frame: At 3, 4 and 6 years of age
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 122 | 129 | 125 | 128
mIU/mL
  anti-HBs; 3 years (N= 118, 130, 122, 119) | 211.1 [147.1 to 303.1] | 189.2 [134.2 to 266.7] | 154.5 [106.8 to 223.5] | 218.9 [152.4 to 314.4]
  anti-HBs; 4 years (N=120, 127, 118, 119) | 130.8 [91.9 to 186.2] | 128.4 [91.3 to 180.6] | 92.3 [63.8 to 133.6] | 142.5 [100.3 to 202.6]
  anti-HBs; 6 years (N=122, 129, 125, 128) | 66.7 [47.2 to 94.1] | 64.7 [46.4 to 90.2] | 45.7 [32.2 to 64.8] | 85.4 [60.4 to 120.6]

34. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 13
Time Frame: From last study contact of the study (NCT00463437) at 17-24 months of age until 6 years of age
Population: Analysis was performed on the Total Enrolled cohort at 6 years of age, which included all subjects vaccinated in the booster study (NCT00463437) and who were part of the blood sample subset.
Measure: Number; unit: Subjects
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Number analyzed (Participants) | 131 | 138 | 135 | 135
Subjects
  SAE(s) | 0 | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From last study contact of the booster study at 17-24 months of age (NCT00463437) until 6 years of age
Description: Since no vaccine was administered during the study, other adverse events were not assessed.
Arm/Group | Synflorix-Meningitec Group | Synflorix-NeisVac-C Group | Synflorix-Menitorix Group | Prevenar-Menitorix Group
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/147 | 0/149 | 0/141
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody when tested by ELISA.The tables show both the results obtained by ELISA and updated results following complete retesting by CLIA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.